CLINICAL TRIAL: NCT03005847
Title: The Effect of Fermented Papaya Preparation on Patients With Chronic Kidney Disease Under Dialysis Receiving Intravenous Iron
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Itamr Sagiv, primary investigator, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FPP001-HMO-CTIL
Record Dates: First submitted 2016-12-26; First posted 2016-12-29 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Anemia; Chronic Kidney Disease Stage 5
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — fermented papaya preparation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FPP arm (Experimental): active treatment with fermented papaya preparation
  Interventions: Dietary Supplement: fermented papaya preparation

INTERVENTIONS:
Dietary Supplement: fermented papaya preparation — dietary supplementation with fermented papaya preparation
  Other Names: FPP

SUMMARY:
Fermented papaya preparation has been reported to bind and neutralize reactive oxygen species as well as iron. Patients undergoing hemodialysis are generally on iron overload status due to their inability to use iron storage adequately. The aim of this study is to evaluate the effect of FPP on the iron status of these patients.

DETAILED DESCRIPTION:
Background and rationale

Patients with chronic kidney disease (CKD) on hemodialysis often suffer from anemia. The anemia is primarily caused by insufficient production by the failing kidneys of the erythroid stimulating hormone - erythropoietin (Epo). Oxidative stress may be another reason for anemia. Oxidative stress in RBCs of these patients may be caused by:

1. Passage of the blood through the plastic tubing during the dialysis procedure. We have shown oxidative stress in RBCs following passage of blood through similar tubing during leukopheresis procedure (1). Other groups reported similar effects during hemodialysis.
2. Iron overload - In order to maximize the effect of Epo, the treatment is supplemented by IV injection of iron. This iron may accumulate and cause iron overload in some hemodialyzed patients. Under normal conditions, iron is transported in the blood and enters into cells following binding the plasma protein transferrin. However, when iron content in the plasma exceeds the binding capacity of transferrin, non-transferrin-bound iron (NTBI) appears. This iron enters cells via alternative pathways, and accumulates in the cytosol, where it participates in chemical reactions (Haber-Weiss, Fenton) that generate reactive oxygen species (ROS). Excess ROS overcomes the protective cellular anti-oxidant mechanisms and becomes cytotoxic. In the erythroid system, excess ROS causes accelerated apoptosis (programmed cell death) of precursor cells in the bone marrow and a short survival of mature RBCs in the circulation, resulting in chronic anemia. Excess iron and ROS may also damage other cells and lead to malfunctioning of vital organs, such as the heart and liver (2,3).

   FPP has been reported to bind and neutralize (scavenge) ROS (4) as well as free iron (chelate) (5). Both activities ameliorate the oxidative stress.

   Treatment with FPP of various diseases associated with oxidative stress, administered orally (3 gr. X 3 times a day), have been shown to significantly ameliorate the symptoms underlying these diseases (6-18). FPP has a long track-record of safe human consumption (19-20). It has been used for many years as a food-supplement by thousands of people around the world without any reported side effect.

   Research goals

   To study the effect of fermented papaya preparation (FPP) on patients with chronic kidney disease (CKD) under dialysis, receiving intravenous iron.

   General Protocol:

   This will be a single-arm, open-label, single-center study in 20 patients upon dialysis receiving IV iron supplementation. All participants will be treated with FPP for 3 months.

   Bi-weekly, blood samples will be drawn and the patients will be monitored for assessment of safety and efficacy.

   Detailed Protocol Twenty patients, treated on Hadassah Medical center, Jerusalem, will be screened and recruited according to clinical criteria.

   inclusion criteria: Age 18-70. Any primary kidney disease resulting in ESRD. Hemodynamically stable status. PTH up to 2-9 times upper normal limits. Patients receiving ESA may be included.
3. Exclusion criteria:

Any evidence of acute bleeding. Hg level of less than 8 g/dL Patients with known allergy to Papaya

3. Patients will be treated orally with FPP (3 gr. X 3 times a day) for 3 months.

4. Blood samples will be obtained from all patients prior and during (every 2 weeks) treatment.

5. Samples will be analyzed for:

Blood chemistry for Potassium, Albumin and Phosphorous (every 2 weeks).

Anemia: Complete blood count, including RBC number and indexes, as well as hemoglobin content.

Oxidative stress: (once monthly) Reactive oxygen species Reduced glutathione Membrane lipid peroxidation External phosphatidylserine

Iron overload: (once monthly) Serum ferritin Serum transferin. Labile plasma iron Serum hepcidin Intracellular labile iron pool

Safety measures:

Adverse events: Frequency, severity, seriousness, time to onset, duration, and relatedness to study product.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70. Any primary kidney disease resulting in ESRD. Hemodynamically stable status. PTH up to 2-9 times upper normal limits. Patients receiving ESA may be included.

Exclusion Criteria:

* Any evidence of acute bleeding. Hg level of less than 8 g/dL Patients with known allergy to Papaya

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Iron status | 3 months of treatment
  evaluation of iron overload reduction after 3 months of treatment with fermented papaya preparation

CONTACTS AND LOCATIONS:
Overall Officials: itamar sagiv, MD, Principal Investigator — Hadassah Medical Organization

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amer J, Frankenburg S, Fibach E. Apheresis induces oxidative stress in blood cells. Ther Apher Dial. 2010 Apr;14(2):166-71. doi: 10.1111/j.1744-9987.2009.00746.x. PMID 20438538
- [Background] Ghoti H, Rachmilewitz EA, Simon-Lopez R, Gaber R, Katzir Z, Konen E, Kushnir T, Girelli D, Campostrini N, Fibach E, Goitein O. Evidence for tissue iron overload in long-term hemodialysis patients and the impact of withdrawing parenteral iron. Eur J Haematol. 2012 Jul;89(1):87-93. doi: 10.1111/j.1600-0609.2012.01783.x. Epub 2012 May 18. PMID 22435497
- [Background] Gaweda AE, Ginzburg YZ, Chait Y, Germain MJ, Aronoff GR, Rachmilewitz E. Iron dosing in kidney disease: inconsistency of evidence and clinical practice. Nephrol Dial Transplant. 2015 Feb;30(2):187-96. doi: 10.1093/ndt/gfu104. Epub 2014 May 12. PMID 24821751
- [Background] Amer J, Goldfarb A, Rachmilewitz EA, Fibach E. Fermented papaya preparation as redox regulator in blood cells of beta-thalassemic mice and patients. Phytother Res. 2008 Jun;22(6):820-8. doi: 10.1002/ptr.2379. PMID 18384199
- [Background] Prus E, Fibach E. The antioxidant effect of fermented papaya preparation involves iron chelation. J Biol Regul Homeost Agents. 2012 Apr-Jun;26(2):203-10. PMID 22824747
- [Background] Bertuccelli G, Marotta F, Zerbinati N, Cabeca A, He F, Jain S, Lorenzetti A, Yadav H, Milazzo M, Calabrese F, Tomella C, Catanzaro R. Iron supplementation in young iron-deficient females causes gastrointestinal redox imbalance: protective effect of a fermented nutraceutical. J Biol Regul Homeost Agents. 2014 Jan-Mar;28(1):53-63. PMID 24750791
- [Background] Marotta F, Naito Y, Jain S, Lorenzetti A, Soresi V, Kumari A, Carrera Bastos P, Tomella C, Yadav H. Is there a potential application of a fermented nutraceutical in acute respiratory illnesses? An in-vivo placebo-controlled, cross-over clinical study in different age groups of healthy subjects. J Biol Regul Homeost Agents. 2012 Apr-Jun;26(2):285-94. PMID 22824755
- [Background] Somanah J, Aruoma OI, Gunness TK, Kowelssur S, Dambala V, Murad F, Googoolye K, Daus D, Indelicato J, Bourdon E, Bahorun T. Effects of a short term supplementation of a fermented papaya preparation on biomarkers of diabetes mellitus in a randomized Mauritian population. Prev Med. 2012 May;54 Suppl:S90-7. doi: 10.1016/j.ypmed.2012.01.014. Epub 2012 Feb 11. PMID 22330753
- [Background] Marotta F, Chui DH, Jain S, Polimeni A, Koike K, Zhou L, Lorenzetti A, Shimizu H, Yang H. Effect of a fermented nutraceutical on thioredoxin level and TNF-alpha signalling in cirrhotic patients. J Biol Regul Homeost Agents. 2011 Jan-Mar;25(1):37-45. PMID 21382272
- [Background] Ghoti H, Fibach E, Dana M, Abu Shaban M, Jeadi H, Braester A, Matas Z, Rachmilewitz E. Oxidative stress contributes to hemolysis in patients with hereditary spherocytosis and can be ameliorated by fermented papaya preparation. Ann Hematol. 2011 May;90(5):509-13. doi: 10.1007/s00277-010-1110-2. Epub 2010 Nov 10. PMID 21063708
- [Background] Aruoma OI, Hayashi Y, Marotta F, Mantello P, Rachmilewitz E, Montagnier L. Applications and bioefficacy of the functional food supplement fermented papaya preparation. Toxicology. 2010 Nov 28;278(1):6-16. doi: 10.1016/j.tox.2010.09.006. Epub 2010 Sep 24. PMID 20870007
- [Background] Marotta F, Koike K, Lorenzetti A, Jain S, Signorelli P, Metugriachuk Y, Mantello P, Locorotondo N. Regulating redox balance gene expression in healthy individuals by nutraceuticals: a pilot study. Rejuvenation Res. 2010 Apr-Jun;13(2-3):175-8. doi: 10.1089/rej.2009.0950. PMID 20370494
- [Background] Fibach E, Tan ES, Jamuar S, Ng I, Amer J, Rachmilewitz EA. Amelioration of oxidative stress in red blood cells from patients with beta-thalassemia major and intermedia and E-beta-thalassemia following administration of a fermented papaya preparation. Phytother Res. 2010 Sep;24(9):1334-8. doi: 10.1002/ptr.3116. PMID 20127662
- [Background] Ghoti H, Rosenbaum H, Fibach E, Rachmilewitz EA. Decreased hemolysis following administration of antioxidant-fermented papaya preparation (FPP) to a patient with PNH. Ann Hematol. 2010 Apr;89(4):429-30. doi: 10.1007/s00277-009-0821-8. Epub 2009 Sep 15. No abstract available. PMID 19756600
- [Background] Marotta F, Yoshida C, Barreto R, Naito Y, Packer L. Oxidative-inflammatory damage in cirrhosis: effect of vitamin E and a fermented papaya preparation. J Gastroenterol Hepatol. 2007 May;22(5):697-703. doi: 10.1111/j.1440-1746.2007.04937.x. PMID 17444858
- [Background] Danese C, Esposito D, D'Alfonso V, Cirene M, Ambrosino M, Colotto M. Plasma glucose level decreases as collateral effect of fermented papaya preparation use. Clin Ter. 2006 May-Jun;157(3):195-8. PMID 16900843
- [Background] Marotta F, Weksler M, Naito Y, Yoshida C, Yoshioka M, Marandola P. Nutraceutical supplementation: effect of a fermented papaya preparation on redox status and DNA damage in healthy elderly individuals and relationship with GSTM1 genotype: a randomized, placebo-controlled, cross-over study. Ann N Y Acad Sci. 2006 May;1067:400-7. doi: 10.1196/annals.1354.057. PMID 16804018
- [Background] Marotta F, Barreto R, Tajiri H, Bertuccelli J, Safran P, Yoshida C, Fesce E. The aging/precancerous gastric mucosa: a pilot nutraceutical trial. Ann N Y Acad Sci. 2004 Jun;1019:195-9. doi: 10.1196/annals.1297.031. PMID 15247013
- [Background] Marotta F, Koike K, Lorenzetti A, Naito Y, Fayet F, Shimizu H, Marandola P. Nutraceutical strategy in aging: targeting heat shock protein and inflammatory profile through understanding interleukin-6 polymorphism. Ann N Y Acad Sci. 2007 Nov;1119:196-202. doi: 10.1196/annals.1404.011. PMID 18056967